CLINICAL TRIAL: NCT06309121
Title: Effects of the Postbiotic Blend ABB C3 on Adiposity and Glucose Metabolism in Children and Adolescents
Acronym: PostOb
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PIC-11-24
Record Dates: First submitted 2024-02-27; First posted 2024-03-13 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Obesity, Childhood; Obesity, Adolescent
Keywords: Obesity; Postbiotics
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Intervention Model Description: Randomized double-blind placebo-controlled study with a treatment group and an active control parallel group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active control (Placebo Comparator): Participants in this arm will receive the usual treatment for obesity at our hospital, based on lifestyle changes (encouraging a healthy diet and physical activity) for 3 months. Participants will receive a daily dose of placebo for these 3 months, then given the option to receive a daily dose of probiotic ABB C3 for 3 more months.
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Follow-up Postbiotic ABB C3 (Optional)
- Treatment (Experimental): Participants in this arm will receive the usual treatment for obesity at our hospital, based on lifestyle changes (encouraging a healthy diet and physical activity) for 3 months. Participants will receive a daily dose of postbiotic blend (ABB C3) for these 3 months, then given the option to receive a daily dose of probiotic ABB C3 for 3 more months.
  Interventions: Dietary Supplement: Postbiotic ABB C3; Dietary Supplement: Follow-up Postbiotic ABB C3 (Optional)

INTERVENTIONS:
Dietary Supplement: Postbiotic ABB C3 — A daily dose of 550 mg of the postbiotic blend ABB C3 in individual sachets for the first 3 months of the study.
  Arms: Treatment
Dietary Supplement: Placebo — A daily dose of 550 mg of the placebo in individual sachets for the first 3 months of the study.
  Arms: Active control
Dietary Supplement: Follow-up Postbiotic ABB C3 (Optional) — Option given to all participants: a daily dose of 550 mg of the postbiotic blend ABB C3 in individual sachets for months 4 to 6 of the study.

SUMMARY:
This study investigates the effects of a postbiotic combination called ABB C3 on reducing body fat and improving metabolic health in children and teenagers. The study consists of a 3-month trial with half participants taking ABB C3 and the other half a placebo, monitoring body composition and blood markers. Afterward, participants can continue with ABB C3 for an additional 3 months. The goal is to determine if ABB C3 is a safe and effective way to help young people improve their health by reducing body fat.

DETAILED DESCRIPTION:
The study focuses on evaluating the effects of a combination of postbiotics called ABB C3 in reducing body fat and improving glucose metabolism. The study proposes a randomized, double-blind clinical trial with participants (aged 8-18 years) randomized into the ABB C3 supplement group or a placebo group. Over a period of 3 months, body composition and relevant blood parameters will be monitored (Study Phase). Subsequently, all participants will be offered to continue with the ABB C3 supplement for an additional 3 months, constituting the Follow-up Phase. The study protocol includes collecting data on possible adverse events. Blood samples and DXA scans will be performed to assess changes in body composition and metabolic health parameters. In summary, the study aims to determine the efficacy and safety of the ABB C3 postbiotic in helping reduce body fat and improve metabolic profiles in children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Age between 8- and 18-year-old
* Obesity (BMI-SDS > 2)

Exclusion Criteria:

* Antibiotic or pre/pro/postbiotic consumption 2 - 4 weeks prior to starting the study
* Chronic diseases affecting glucose or lipid metabolism
* Chronic medication affecting glucose or lipid metabolism, or inducing a pro-inflammatory state
* History of bariatric surgery
* Diabetes requiring insulin treatment
* Severe intellectual disability
* Pregnancy
* Individuals taking medications that may alter appetite or weight, with a recent change in prescription within the last 3 months or anticipated changes during the 2 months of participation

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | Baseline, 1.5 months, 3 months
  Treatment safety and tolerability will be evaluated by assessing differences in the incidence of potential adverse events between groups, focusing on gastrointestinal symptoms.
Change in adiposity (% fat body mass) | 3 months
  Fat body mass (adiposity) will be assessed by dual energy x-ray absorptiometry (DXA) scan at baseline and 3 months and differences will be assessed
Change in blood glycated hemoglobin (HbA1c) levels | 3 months
  Blood tests will be performed at baseline and 3 months and HbA1c (%) levels quantified.

SECONDARY OUTCOMES:
Change in adiposity (% fat body mass) | Baseline, 6 months
  Fat body mass (adiposity) will be assessed by dual energy x-ray absorptiometry (DXA) scan at baseline and 6 months and differences will be assessed.
Change in blood glycated hemoglobin (HbA1c) levels | Baseline, 6 months
  Blood tests will be performed at baseline and 6 months and HbA1c (%) levels quantified. Differences between time-points will be assessed.
Change in BMI z-score | Baseline, 1.5 months, 3 months, 6 months
  Weight and height will be combined to calculate changes in BMI and BMI z scores and differences between time-points will be assessed.
Change in body composition | Baseline, 1.5 months, 3 months, 6 months
  Body composition (lean and fat mass) will be estimated by bioimpedance and differences between time-points will be assessed.
Change in insulin sensitivity | Baseline, 3 months, 6 months
  Fasting blood glucose and insulin concentrations will be combined to calculate HOMA-IR (Homeostatic Model Assessment for Insulin Resistance) and differences between time-points will be assessed
Change in lipid profile (triglycerides, cholesterol) | Baseline, 3 months, 6 months
  The lipid profile will be determined by blood test and differences between time-points will be assessed
Change in blood pressure | Baseline, 3 months, 6 months
  Both systolic and diastolic blood pressure will be measured at each visit and differences between time-points will be assessed
Change in Beck Depression Inventory-II (BDI-2) | Baseline, 3 months, 6 months
  The Beck Depression Inventory for Youth (BDI-2) assesses negative thoughts of children or adolescents about themselves, their life, and their future, along with feelings of sadness and physiological signs of depression. It is a 20-item questionnaire with a score range of 0-60. Higher scores indicate worse outcome.
Change in Beck Anxiety Inventory-II (BAI-2) | Baseline, 3 months, 6 months
  The Beck Anxiety Inventory for Youth (BAI-2) assesses the fears and concerns of children or adolescents, as well as physical symptoms associated with anxiety. It is a 20-item questionnaire with a score range of 0-60. Higher scores indicate worse outcome.

OTHER OUTCOMES:
Change in gut microbial abundance and diversity | Baseline, 3 months, 6 months
  DNA will be isolated from fecal samples and analyzed by deep-sequencing to determine the composition, abundance, and diversity of gut microbiota.
Change in plasma metabolite concentrations | Baseline, 3 months, 6 months
  Metabolite concentrations in plasma samples will be measured by liquid chromatography coupled to mass spectrometry (metabolomics).

CONTACTS AND LOCATIONS:
Overall Officials: Carles Lerin, PhD, Principal Investigator — Fundació Sant Joan de Deu
Locations (1):
- Hospital Sant Joan de Déu, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No